CLINICAL TRIAL: NCT01549717
Title: Feasibility And Efficacy Of Continuous In-Hospital Patient Monitoring
Acronym: LISTEN
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Guy's and St Thomas' NHS Foundation Trust (Other)
Collaborators: Engineering and Physical Sciences Research Council, UK (Other); King's College London (Other); University of Oxford (Other)
Responsible Party: Principal Investigator, Richard Beale, Consultant, Guy's and St Thomas' NHS Foundation Trust
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 12/LO/0526
Record Dates: First submitted 2012-03-07; First posted 2012-03-09 (Estimated); Last update posted 2014-02-12 (Estimated); Status verified 2014-02

CONDITIONS: Monitoring of Patients Following Surgery
Keywords: Early warning score; Physiological score; Track and trigger score; Scoring system; Physiological model; Monitoring; Patient monitoring; Wireless monitoring; Wearable monitor

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Elective cardiac surgery patients (Experimental): Patients undergoing elective cardiac surgery
  Interventions: Device: Fitting of a wireless telemetry device

INTERVENTIONS:
Device: Fitting of a wireless telemetry device — Fitting of a Philips Intellivue Trx + SpO2 telemetry device. To be worn throughout patient stay except if being monitored using a standard bedside monitor or bathing.
  Other Names: Philips Intellivue Trx + SpO2

SUMMARY:
The investigators plan to study patients who have had cardiac surgery. Current standard practice is to monitor patients who have had cardiac surgery using wall-mounted monitors whilst they are on the Overnight Intensive Recovery (OIR) and the cardiac High Dependency Unit (HDU). The wall-mounted monitors monitor the vital signs continuously and alert the nurses if any abnormalities are detected. Once a patient is transferred from HDU to the cardiac surgery ward for the most part they are no longer connected to a continuous monitor. Instead, the majority of patients on the ward have their vital signs only intermittently checked during the day, using a "spot check monitor". There is a small minority, chosen on clinical grounds, who are assessed with wireless "telemetry" monitors for a day or two.

In this study the investigators will continuously monitor the vital signs of all enrolled patients from the time that they leave the operating theatre to the the time they are discharged from hospital. Whilst they are on OIR and HDU they will be monitored with the standard wall-mounted monitors in the normal fashion. When they then move to the ward the investigators will give all enrolled patients a telemetry monitor to wear as well as asking the nurses to check their vital signs with spot check monitors.

The investigators will also collect information about the patients' general state of health and record indicators of worsening in patients' condition so that the investigators can determine how changes in the vital signs relate to deterioration. Finally the investigators plan to survey the patients and nurses to understand their experiences of continuous monitoring and what needs to be changed to improve the patient experience.

ELIGIBILITY:
Inclusion Criteria:

* Adult (aged over 18 years old)
* Planned for elective cardiac surgery
* Post surgery care is planned to be on a study ward

Exclusion Criteria:

* Inability or refusal to consent
* Pregnant
* Prisoners
* For palliative care only

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2012-12; Primary Completion 2014-02 (Actual); Study Completion 2014-02 (Actual)

PRIMARY OUTCOMES:
The number of patients in whom abnormal vital signs are detected by a continuous monitor more than an hour before they are detected according to standard ward practice

SECONDARY OUTCOMES:
The proportion of patient stay for which good quality continuous data is captured
The number of alerts caused by probe off alarms and artefactual readings
The sensitivity of the automated early warning score developed from this data for predicting clinical deterioration
The specificity of the automated early warning score developed from this data for predicting clinical deterioration

CONTACTS AND LOCATIONS:
Overall Officials: Richard Beale, MBBS, Principal Investigator — Guy's & St Thomas' Foundation Trust
Locations (1):
- St Thomas' Hospital, London, London, United Kingdom